CLINICAL TRIAL: NCT01968148
Title: Mechanisms of Ultra-acute Hyperglycemia After Successful Resuscitation From Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jouni Nurmi, MD, MD, PhD, Helsinki University Central Hospital
Other Study IDs: 357/13/03/12/2012 § 205
Record Dates: First submitted 2013-10-19; First posted 2013-10-23 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Heart Arrest; Cardiac Arrest
Keywords: glucose; cardiac arrest; resuscitation; insulin; GLP-1
MeSH Terms: conditions — Heart Arrest; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to describe the mechanisms of ultra-acute hyperglycemic response after return of spontaneous circulation (ROSC) in patients suffering out-of-hospital cardiac arrest. The investigators hypothesize that ischemia and reperfusion injury leads decreased secretion of insulin and glucose-like peptide 1 (GLP-1).

Two blood samples will be drawn: (1.) Immediately after ROSC and (2.) 60 minutes after first sample. Concentrations of glucose, insulin, glucagon and GLP-1 will be compared between the samples.

Metabolic profile will be compared between: (1.) diabetic and non-diabetic patients and (2.) survivors and non-survivors.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* witnessed cardiac arrest
* interval form emergency call to return of spontaneous circulation 10-45 minutes

Exclusion Criteria:

* severe pre-arrest disability leading to withdrawing treatment in prehospital phase
* no concent from next of kin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Successfully resuscitated patients treated by physician staffed mobile intensive care unit in Helsinki area.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Change in level of insulin | 60 minutes
Change in level of glucagon | 60 minutes

SECONDARY OUTCOMES:
Blood cortisol level | 60 minutes after ROSC
Blood interleukin-6 level | 60 minutes after ROSC
Change in blood glucose level | 60 minutes
Change in level of GLP-1 | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jouni Nurmi, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki Emergency Medical Services, Helsinki
  - Helsinki Area Helicopter Emergency Medical Services, Vantaa